CLINICAL TRIAL: NCT06581211
Title: Aromatherapy Oil Associated Changes on Anxiety and Pain During Bone Marrow Biopsy Procedures
Brief Title: Aromatherapy Oil Associated for Managing Anxiety and Pain During Bone Marrow Biopsy Procedures
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual goal met
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23234; P30CA033572 (NIH); NCI-2024-05514 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23234 (Other: City of Hope Medical Center)
Record Dates: First submitted 2024-07-16; First posted 2024-09-03 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Aromatherapy; jojoba wax; lavender oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (LOA) (Experimental): Patients inhale LOA for 20 minutes prior to SOC BMAB and throughout the procedure.
  Interventions: Other: Electronic Health Record Review; Other: Lavender Oil; Other: Questionnaire Administration
- Group II (LA) (Experimental): GROUP II: Patients inhale LA for 20 minutes prior to SOC BMAB and throughout the procedure.
  Interventions: Procedure: Aromatherapy and Essential Oils; Other: Electronic Health Record Review; Other: Questionnaire Administration
- Group III (jojoba) (Placebo Comparator): Patients inhale jojoba oil for 20 minutes prior to SOC BMAB.
  Interventions: Other: Electronic Health Record Review; Other: Jojoba Oil; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Aromatherapy and Essential Oils — Inhale LA
  Other Names: Aromatherapy
  Arms: Group II (LA)
Other: Electronic Health Record Review — Ancillary studies
Other: Jojoba Oil — Inhale jojoba oil aromatherapy
  Arms: Group III (jojoba)
Other: Lavender Oil — Inhale LAO
  Other Names: Common Lavender Oil; English Lavender Oil; Lavandula officinalis Flowering Top Oil
  Arms: Group I (LOA)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates whether using aromatherapy can reduce pain and anxiety for cancer patients during routine biopsy procedures. Because of the discomfort associated with a bone marrow aspirate and biopsy (BMAB), many patients have significant anxiety in addition to their pain. With the current background of the opioid crisis, researchers have been looking for different ways to treat pain and anxiety in cancer patients without using medications that have a risk for abuse. Recent research suggests that using lavender aromatherapy may be an effective and more affordable treatment for anxiety and pain in patients. Information gathered from this study may help researchers determine whether using aromatherapy may help to manage pain and anxiety during biopsy procedures for cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of utilizing aromatherapy oils during bone marrow biopsy procedures in clinical practice.

II. To assess satisfaction of patients receiving aromatherapy oils during bone marrow biopsy procedures in clinical practice.

SECONDARY OBJECTIVES:

I. To observe the relationship of aromatherapy oils (as compared to placebo aromatherapy) on anxiety in patients undergoing a bone marrow aspirate and biopsy procedure.

II. To observe the relationship of aromatherapy oils (as compared to placebo aromatherapy) on pain in patients undergoing a bone marrow aspirate and biopsy procedure.

III. To observe the relationship of aromatherapy oils (versus placebo aromatherapy) on other symptoms (i.e., physical, emotional symptoms, etc.).

IV. Additionally assess if there are any differences in practitioner procedure evaluation between the groups.

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP I: Patients inhale lavender oil aromatherapy (LAO) for 20 minutes prior to standard of care (SOC) BMAB and throughout the procedure.

GROUP II: Patients inhale linalool oil aromatherapy (LA) for 20 minutes prior to SOC BMAB and throughout the procedure.

GROUP III: Patients inhale jojoba oil aromatherapy for 20 minutes prior to SOC BMAB.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and sign a written informed consent document, and be willing to follow protocol requirements
* Ability to read and understand English for patient reported outcomes
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Willingness to comply with all study interventions of essential oil aromatherapy
* Anxiety > 3 on a 0-10 visual analog scale regarding the bone marrow biopsy/aspirate procedure
* The study is open to all participants regardless of gender, race, or ethnicity

Exclusion Criteria:

* Allergy to lavender oil, linalool oil, jojoba oil
* Previous enrollment in this study
* Uncontrolled respiratory conditions such as asthma and chronic obstructive pulmonary disease (COPD)
* Mental incapacitation (ex. stroke, brain metastasis etc.) that would cause inability to follow directions, in the opinion of the investigators
* Ongoing uncontrolled active psychiatric condition that would interfere in the conduct of the study (e.g., mood disorders, anxiety, psychosis disorders, or substance use), as determined by the patient's primary cancer team.

  * If a patient has a history of a psychiatric disorder, we will contact their primary cancer team to determine if their condition is controlled or uncontrolled, and if it will interfere with the study
* Recent changes in the past 2 weeks to medications prescribed for pain or anxiety
* Abnormal smelling abilities due to sinus infections, long COVID, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients participated in the aromatherapy oils (Feasibility) | Up to 1 month
  Will consider the study feasible if > 70% of patients are able to complete the oil treatment (lavender, linalool or placebo). Will be estimated within 95% confidence interval.
Proportion of patients completed the aromatherapy oils (Feasibility) | Up to 1 month
  Completion will be defined as receiving oil treatments as described. Each patient will be assigned one of the following categories: 1) complete treatment course, 2) incomplete treatment course, or 3) unknown (not assessable, insufficient data). Will be estimated within 95% confidence interval.
Patient satisfaction | One time patient satisfaction assessment within 30 minutes after bone marrow aspiration and biopsy (BMAB).
  Will be evaluated using a survey, in order to fully understand their experience with the treatment. Will also evaluate whether the patients are interested in aromatherapy oils for future bone marrow aspiration and biopsy (BMAB), and their experience in the clinical trial. Descriptive analyses (exploratory) will be provided for all individual assessment items.

SECONDARY OUTCOMES:
Association between aromatherapy and other symptoms | The 3 time points are: at baseline before oil administration; after oil administration before BMAB; after BMAB up to 24 hours
  Will be compared (to placebo aromatherapy) using the ESAS scores for the remaining symptoms via the mixed effect modeling approach. For individual scores, research indicates a change of 1.0-1.5 correlates with a minimal clinically important difference.
Association between aromatherapy and anxiety | The 3 time points are: at baseline before oil administration; after oil administration before BMAB; after BMAB up to 24 hours
  We will compare differences in anxiety scores between each intervention aromatherapy group (Lavender, Linalool) and Placebo (Jojoba) using independent sample t-test (or Mann-Whitney test). We will assess anxiety scores from the ESAS form, within and between groups, at three specific assessment points (pre-BMAB, post-relaxation, and post-BMAB) via mixed effect regression models (which will account for the correlation between observations on the same patient). We will test for time, and group by time interaction effects.
Clinician's responses | At post-BMAB up to 24 hours
  Will be assessed using the post-procedure questionnaire. Descriptive analyses will be produced (by group). Furthermore, independent samples t-tests will be applied to determine if there are any differences in practitioner procedure evaluation questions between the two groups.
Association between aromatherapy and pain | The 3 time points are: at baseline before oil administration; after oil administration before BMAB; after BMAB up to 24 hours
  Will be compared (to placebo aromatherapy) using scores from the pain question of the ESAS. Will also use the Brief Pain Inventory Short Form total score. A statistical analysis similar to the comparison in anxiety scores will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Lee, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Lennar, Irvine, California